CLINICAL TRIAL: NCT00561483
Title: Sequential Cystatin C Levels and Renal Impairment in Acute Heart Failure
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wilson Tang, Principal Investigator, staff cellular and molecular medicine and cardiovascular medicine, The Cleveland Clinic
Other Study IDs: 07-834
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Acute Heart Failure; Renal Failure
Keywords: Acute heart failure; cystatin C; renal failure; biomarker
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients admitted to the hospital with decompensated heart failure

SUMMARY:
Renal Compromise after treatment of decompensated heart failure with diuretics is not uncommon. The purpose of our study is to investigate the relationship between cystatin C and worsening renal function in this setting. Cystatin C is a biomarker produced at a constant rate by all cells that is a sensitive biomarker of renal function.Cystatin C and Plasma amino terminal proB-type natriuretic peptide (NT-proBNP) levels will be obtained at baseline and daily. Our goal is to enroll 100 subjects with an estimated 5 samples per each subject. The time course of changes in cystatin C in relation to serum creatinine levels over time will be plotted.

Our hypothesis is that sequential changes in cystatin C levels following initial treatment with diuretic therapy in the setting of acute decompensated heart failure may provide early insight into cardio-renal compromise. Understanding the natural history and time course of the changes in sequential cystatin C levels may facilitate further studies to guide the judicious use of diuretic therapy in acute decompensated heart failure, and to predict the risk of subsequent development of worsening renal function. If serial testing of cystatin C can provide accurate assessment and prediction of worsening renal function, clinical applications of these observations can be evaluated in future prospective studies.

DETAILED DESCRIPTION:
This is a single-center, prospective, cohort study. The design of this pilot study focuses on the feasibility to complete the project in a short period of time by the applicant. Subjects will be identified in the morning after their hospital admission and informed consent will be obtained for the study. At the time of enrollment blood samples and urine samples will be collected as baseline, together with a brief history and physical examination to document degree of congestion and basic vital signs. In addition their unused (to be discarded) blood samples from previous clinical labs from this admission may be retrieved from the clinical laboratory.

Patients will be followed daily, and each day a blood draw and urine sample will be obtained for research purposes until the day of discharge. Changes in vital signs, available laboratory data for serum creatinine and BUN, and congestion score will be documented. Physicians treating the patient will be blinded from the laboratory results. Because of the small sample size and the low anticipated rate of adverse events, this study uses a combined outcome of either death in hospital, death within 90 days after discharge or readmission to the hospital facility for heart failure within 90 days. Patients will be called after 90 days for follow up if readmission or death information is not available in the Electronic Medical Record.

Specific aims include:

Specific Aim 1 - To examine the natural history of changes in sequential cystatin C levels during diuretic therapy in Acute Decompensated Heart Failure.

Specific Aim 2 - To determine the predictive value of changes in sequential cystatin C levels to subsequent development of worsening renal function (WRF) and WRF in association with aminoterminal pro B-type natriuretic peptide (NT-proBNP) levels.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission within 48 hours for ADHF, with an expected stay over 24 hours.
* Evidence of fluid overload, including jugular venous distention, pulmonary rales, peripheral edema, and/or ascites receiving diuretic therapy

Exclusion Criteria:

* Heart failure due to congenital heart disease or critical aortic stenosis (potentially different cardio-renal pathophysiology)
* Acute myocardial infarction or unstable acute coronary syndromes
* End-stage renal insufficiency on renal replacement therapy (already has underlying advanced renal failure).
* Patients with active cancer (cystatin C has been shown to be produced by some tumors)
* Known exposure to nephrotoxic agents (such as contrast dye) or planned surgery during hospitalization at the time of enrollment
* Hemoglobin < 9 mg/dL or clinically significant active bleeding.
* Unable to comply with protocol or unable to have informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital with decompensated heart failure
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2007-12-05 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
To examine the natural history of cystatin C levels during diuretic therapy in ADHF | 7 days
  To examine the natural history of cystatin C levels during diuretic therapy in ADHF

SECONDARY OUTCOMES:
To determine the predictive value of changes in sequential cystatin C levels to subsequent development of WRF | 7 days
  To examine the natural history of cystatin C levels during diuretic therapy in ADHF
The combined outcome of either death in hospital or death within 90 days after discharge or readmission to the hospital facility for heart failure within 90 days | 90 days
  The combined outcome of either death in hospital or death within 90 days after discharge or readmission to the hospital facility for heart failure within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: W. H. Wilson Tang, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No